CLINICAL TRIAL: NCT05829109
Title: Safety and Efficacy of Healthy to Inflamed Pouch Fecal Microbiota Transplantation
Brief Title: Fecal Microbiota Transplant for Patients With Chronic Pouchitis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Maia Kayal (Other)
Responsible Party: Sponsor-Investigator, Maia Kayal, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-01753
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pouchitis; Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This will be a pilot study of 16-18 patients who will each receive FMT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fecal Microbiota Transplant (FMT) (Experimental): Single arm of 16-18 subjects, all of whom will receive the interventional FMT.
  Interventions: Drug: Fecal Microbiota Transplant (FMT)

INTERVENTIONS:
Drug: Fecal Microbiota Transplant (FMT) — The intervention consists of the following steps:
  * Step 1: Vancomycin 125 mg orally every 6 hours and metronidazole 250 mg orally every 6 hours for 5 days.
  * Step 2: Bowel preparation with 10 ounces of magnesium citrate.
  * Step 3: Two FMT doses will be administered via enema one week apart using stool from donors with a durably healthy pouch.

SUMMARY:
The purpose of this research study is to assess the safety and efficacy of fecal microbiota transplant (FMT) in the treatment of chronic pouchitis.

DETAILED DESCRIPTION:
The purpose of this research study is to assess the safety and efficacy of fecal microbiota transplant (FMT) in the treatment of chronic pouchitis. FMT has been successfully used in the treatment of recurrent Clostridiodes difficile infection and has shown benefit in the treatment of ulcerative colitis in clinical trials. The success of FMT in these patients is because of the reconstitution of the recipient's unhealthy gut bacteria with the donor's healthy gut bacteria.

Surgery to remove the colon is required in a subset of patients with ulcerative colitis that does not respond to medical therapy. In these patients, an internal pouch is created from small intestine to function as a stool reservoir and avoid an ostomy after the colon is removed. Inflammation of the pouch, pouchitis, is common after surgery and can manifest as diarrhea, pelvic pain, urgency and blood in the stool. Chronic pouchitis occurs in up to 20% of patients and there is no approved treatment. A number of studies have evaluated FMT in patients with chronic pouchitis, but have proven unsuccessful. This is likely because these studies have used stool from patients with a colon and transplanted it into patients with a pouch. This is problematic because the gut bacteria of the colon and pouch are not similar, and putting healthy stool from a colon may not reconstitute a healthy pouch microbiome. The specific purpose of this project is to transplant stool from patients with a healthy pouch to patients with an inflamed pouch.

ELIGIBILITY:
Inclusion Criteria:

Patients age 18 or greater with UC who have undergone TPC with IPAA and have one of the following chronic pouchitis phenotypes, each defined as:

* Chronic antibiotic dependent pouchitis:
* The need for continuous antibiotic therapy (>4 weeks) to maintain clinical remission and a history of at least 2 attempts in the last 24 months to stop antibiotic therapy resulting in pouchitis episodes, OR
* Active pouchitis with a modified Pouchitis Disease Activity Index (mPDAI) ≥5 and a history of ≥4 antibiotic therapies in the last 12 months
* Chronic antibiotic refractory pouchitis:
* Active pouchitis with a modified Pouchitis Disease Activity Index (mPDAI) ≥5 with no response to antibiotics
* Crohn's disease like pouch inflammation on biologic or small molecule therapy with persistent symptoms:
* Pre-pouch ileal inflammation, strictures, and/or fistulae, AND
* Active biologic or small molecule therapy, AND
* Persistent symptoms with mPDAI clinical sub-score ≥ 2

Exclusion Criteria:

Patients with UC who underwent TPC with IPAA and meet one of the following criteria will be excluded:

* Allergy to vancomycin, metronidazole, or ingredients present in the FMT
* Women who are breastfeeding
* Women who are pregnant
* Participants with fever > 100.4F/38C or other signs of active illness
* Active treatment with biologics (infliximab, adalimumab, golimumab, vedolizumab, ustekinumab)
* Active treatment with immunomodulators (azathioprine, 6-mercaptopurine, methotrexate), steroids or any investigational drugs
* Crohn's disease like pouch inflammation
* Active enteric infection
* Isolated cuffitis
* Clinically significant strictures of the pouch inlet or outlet
* Participation in a clinical trial in the preceding 30 days
* Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines will put the participant at greater risk from FMT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with FMT related adverse events | 8 weeks
  The number of patients with FMT related adverse events through week 8 classified according to the Medical Dictionary for Regulatory Activities (MedDRA) and categorized according to the NIH Criteria for Adverse Events.

SECONDARY OUTCOMES:
Number of patients in clinical remission | 8 weeks
  The number of patients in clinical remission assessed via patient interview and defined as mPDAI clinical subscore ≤4 points and no need for antibiotic therapy at week 8.
Number of patients with endoscopic response | 8 weeks
  The number of patients with endoscopic response assessed via pouchoscopy and defined as a decrease from baseline in mPDAI endoscopic subscore > 2 points at week 8.
Change in recipient fecal microbial diversity via metagenomics analysis | Baseline and up to 8 weeks
  The change in recipient fecal microbial diversity after FMT relative to baseline assessed via stool collection and using metagenomics analysis.
Change in recipient fecal microbial diversity via strain strain isolation | Baseline and up to 8 weeks
  The change in recipient fecal microbial diversity after FMT relative to baseline assessed via strain isolation - to isolate and sequence the gut microbial strains from each donor
Change in recipient microbe tracking | Baseline and up to 8 weeks
  The change in recipient fecal microbial diversity after FMT relative to baseline assessed by recipient microbe tracking.
Change in B cells | Baseline and 8 weeks
  The change in the mucosal immune profile before and after FMT as measured by B cells
Change in myeloid cells | Baseline and 8 weeks
  The change in the mucosal immune profile before and after FMT as measured by myeloid cells
Change in T cells | Baseline and 8 weeks
  The change in the mucosal immune profile before and after FMT as measured by T cells
Change in NK cell subsets | Baseline and 8 weeks
  The change in the mucosal immune profile before and after FMT as measured by NK cell subsets

CONTACTS AND LOCATIONS:
Overall Officials: Maia Kayal, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. For individual participant data meta-analysis. Proposals should be directed to Maia.Kayal@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (tbd).